CLINICAL TRIAL: NCT00139360
Title: Efficacy of Bevacizumab Monotherapy in Treatment of Metastatic Melanoma and Predictive Value of Angiogenic Markers
Brief Title: Efficacy of Bevacizumab Monotherapy in Treatment of Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: Norwegian Cancer Society (Other); Hoffmann-La Roche (Industry)
Responsible Party: Principal Investigator, Oddbjørn Straume, MD PhD, MD PhD, Haukeland University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSD-11933; 94070/013
Record Dates: First submitted 2005-08-30; First posted 2005-08-31 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — Bevacizumab

ARMS (1):
- 1 (Experimental): Active drug
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Anti angiogenesis treatment

SUMMARY:
To determine the efficacy as measured by objective tumor response of first-line treatment of metastatic melanoma with bevacizumab monotherapy

DETAILED DESCRIPTION:
In Norway, cutaneous malignant melanoma is the second most frequent and the most frequent cancer type in middle-aged (30-54 years) females and males, respectively, and the incidence has six-doubled during the last 30 years. Median survival for patients with metastatic melanoma is 6 months.

Many agents have been investigated for anti-tumor effect in melanoma, but there is no accepted standard therapy. Biochemotherapy, combining cytotoxic drugs with Interleukin-2 or Interferon alpha, has not been shown to be superior to single agent Dacarbazine (DTIC), which is regarded to be the most active agent. Other biological approaches like vaccination are currently under investigation, but still no efficient treatment for metastatic melanoma is available. DTIC induces objective remission in 20% of the patients, but without significant impact on survival.

The need of a new and effective treatment for the group of melanoma patients is urgently needed. This will be the first study to assess response rates of bevacizumab monotherapy in first line treatment of metastatic melanoma. In addition there will be a major focus on the identification of predictive biomarkers of bevacizumab efficacy.

ELIGIBILITY:
LEVEL A (second line): after confirmed progression on standard first line treatment with dacarbazine.

LEVEL B (first line): when objective clinical response is observed in LEVEL A, patients will be included for first line treatment with bevacizumab

Inclusion Criteria:

* Histologically confirmed metastatic (unresectable) melanoma and with progressive disease
* WHO performance status 0-2
* Age >18 years
* Able to undergo outpatient treatment
* Patients must have clinically and/or radiographically documented measurable disease according to RECIST criteria
* At least 4 weeks since adjuvant interferon alpha
* Recovered from prior chemotherapy
* Major surgical procedure or significant traumatic injury within 28 days prior to study treatment start. Biopsy or fine needle aspiration within 5 days prior to study treatment start. Central venous line placement must be inserted at least 5 days prior to treatment start.
* Minimum required laboratory data:

Hematology: absolute granulocytes > 1.0 x 109/L platelets > 100 x 109/L Biochemistry: bilirubin < 1.5 x upper normal limit serum creatinine within normal limits INR < 1.5

* Before patient registration/randomization, written informed consent must be given according to national and local regulations.

Exclusion Criteria:

* No pregnant or lactating patients can be included
* No prior interferon alpha or IL-2 for metastatic disease
* No more than 1 prior chemotherapy regimen for metastatic disease
* No clinical evidence of coagulopathy
* No brain metastases
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No history of thrombosis
* No full-dose oral coumarin-derived anticoagulants (INR>1.5) or heparin, thrombolytic agents, or chronic, daily treatment with aspirin (>325 mg/day)
* No non-steroidal anti-inflammatory medications (those known to inhibit platelet function at doses used to treat chronic inflammatory diseases)
* No uncontrolled hypertension
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2005-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Clinical Response rates | Evaluated by CT scans every 12 weeks, later every 6 monts. Up to 10 years.

SECONDARY OUTCOMES:
Time to progression | Evaluated by CT scans every 12 weeks, later every 6 monts. Up to 10 years.
Overall survival | Evaluated by CT scans every 12 weeks, later every 6 monts. Up to 10 years.
Safety data | Evaluated by consultations every 12 weeks, later every 6 monts. Up to 10 years.
  CTCAEv2 side effects

CONTACTS AND LOCATIONS:
Overall Officials: Oddbjorn Straume, MD, PhD, Principal Investigator — Department of Oncology, Haukeland University Hospital
Locations (1):
- Department of Oncology, Haukeland University Hospital, Bergen, Norway

REFERENCES:
- [Derived] Schuster C, Akslen LA, Straume O. Expression of Heat Shock Protein 27 in Melanoma Metastases Is Associated with Overall Response to Bevacizumab Monotherapy: Analyses of Predictive Markers in a Clinical Phase II Study. PLoS One. 2016 May 11;11(5):e0155242. doi: 10.1371/journal.pone.0155242. eCollection 2016. PMID 27166673
- [Derived] Schuster C, Eikesdal HP, Puntervoll H, Geisler J, Geisler S, Heinrich D, Molven A, Lonning PE, Akslen LA, Straume O. Clinical efficacy and safety of bevacizumab monotherapy in patients with metastatic melanoma: predictive importance of induced early hypertension. PLoS One. 2012;7(6):e38364. doi: 10.1371/journal.pone.0038364. Epub 2012 Jun 15. PMID 22719881